CLINICAL TRIAL: NCT00656617
Title: Phase II Study of Idarubicin, Cytarabine, and Vorinostat in Patients With High-Risk MDS and AML
Brief Title: Phase II Study of Idarubicin, Cytarabine, and Vorinostat With High-Risk Myelodysplastic Syndrome (MDS) and Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0835; NCI-2010-01500 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Results first posted 2015-03-09 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-02

CONDITIONS: Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS)
Keywords: Acute Myeloid Leukemia; (AML); Myelodysplastic syndrome; (MDS); Leukemia; Idarubicin; Cytarabine; Vorinostat; Ara-C
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia | interventions — Idarubicin; Cytarabine; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Idarubicin + Ara-C + Vorinostat (Experimental): Idarubicin 12 mg/m^2 by vein (IV) over 1 hour daily for 3 days (days 4 to 6). Ara-C (Cytarabine) 1.5 g/m^2 IV as a continuous infusion over 24 hours daily (days 4 to 7). Vorinostat initial dose level 500 mg orally three times a day for 3 days (days 1 to 3).
  Interventions: Drug: Idarubicin; Drug: Cytarabine; Drug: Vorinostat

INTERVENTIONS:
Drug: Idarubicin — 12 mg/m^2 IV over 1 hour daily for 3 days (days 4 to 6)
  Other Names: Idamycin PFS®
Drug: Cytarabine — 1.5 g/m^2 IV as a continuous infusion over 24 hours daily (days 4 to 7)
  Other Names: Ara-C; Cytosine arabinoside; Cytosar-U®; DepoCyt
Drug: Vorinostat — Initial dose level 500 mg orally three times a day for 3 days (days 1 to 3).
  Other Names: Zolinza®; SAHA; Suberoylanilide Hydroxamic Acid; MSK-390

SUMMARY:
The goal of this clinical research study is to find the highest safe dose of vorinostat that can be given in combination with idarubicin and ara-C for the treatment of AML and high-risk MDS.

Once the highest safe dose is found, researchers will then try to learn if this combination treatment can help to control AML and high-risk MDS in newly diagnosed patients. The safety of this treatment combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Vorinostat is designed to change the gene expression profile of leukemia cells, which may cause the cells to die.

Idarubicin is designed to cause breaks in DNA (the genetic material of cells). This may cause cancer cells to die.

Ara-C is designed to insert itself into DNA of cancer cells and stop the DNA from repairing itself.

This dose combination has not been tested in humans before, at this dose level and schedule.

Study Drug Administration:

Induction Therapy:

If you are found to be eligible to take part in this study, you will begin induction therapy. During induction therapy, the dose level of vorinostat may vary based on when you join the study and on the side effects seen in other participants. The first group of 3 participants will receive the highest dose level of vorinostat. If intolerable side effects are experienced, the next group of 3 participants will receive a lower dose of vorinostat. This will continue until the highest dose of vorinostat with no intolerable side effects is found. The dose levels of the other drugs will not change.

In the Induction phase, you will receive 1 or 2 induction cycles of therapy on the following schedule:

* On Days 1-3, you will take vorinostat by mouth 3 times a day.
* On Days 4-6, you will receive idarubicin through a needle in your vein over 1 hour.
* On Days 4-7, you will receive ara-C by vein as a non-stop infusion.
* On Days 4-7, you will receive solumedrol or dexamethasone to help reduce the risk of side effects associated with ara-C. The drug will be given by vein over a few seconds.

Consolidation Therapy:

If the disease responds during Induction, you may be able to receive up to 5 additional 4-6 week study cycles. During these Consolidation Cycles, you will take the study drugs on the following cycle:

* On Days 1-3, you will take vorinostat by mouth 3 times a day.
* On Days 4 and 5, you will receive idarubicin through a needle in your vein over 5 minutes.
* On Days 4-6, you will receive ara-C by vein as a non-stop infusion.
* On Days 4 and 5, you will also receive either solumedrol or dexamethasone by vein over a few seconds.

Maintenance Therapy:

If you go into remission, you will begin maintenance therapy. While on maintenance therapy, you will take vorinostat by mouth 3 times a day on Days 1-14 of each 28-day study cycle. You may have up to 12 Maintenance Cycles.

Study Visits:

At least every week during Cycle 1, and then at least once a month during each additional cycle, blood (about 1-2 teaspoons) will be drawn for routine tests. You will also have routine bone marrow aspirates and biopsies before initiating treatment and approximately on Day 21 and Day 28 after initiating therapy.

Length of Study:

You may continue to receive the study drugs for up to 18 cycles. You will be taken off study early if the disease gets worse or intolerable side effects occur.

This is an investigational study. Idarubicin is FDA approved for use in combination with other approved drugs for the treatment of AML. Vorinostat is FDA approved and commercially available for the treatment of some forms of cutaneous lymphoma. Ara-C is FDA approved for use in the treatment of leukemia. The use of these drugs together is investigational.

Up to 105 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of 1) AML (World Health Organization (WHO) classification definition of >/= 20% blasts), or 2) intermediate-2 or high-risk MDS (defined by the IPSS classification2).
2. Patients aged 15 to 65 years;
3. For the initial run-in phase of the study, patients with relapsed or refractory disease or patients with secondary untreated disease are eligible, however, these patients must not have had prior exposure to a histone deacetylase inhibitor, prior antecedent hematological disorder or secondary disease with complex cytogenetics.
4. For the actual phase II portion of the study: patients must be chemonaïve, i.e., not have received any chemotherapy (except hydrea) for AML or MDS. They may have received hypomethylating agents for prior MDS and transfusions, hematopoietic growth factors or vitamins. Temporary prior measures such as apheresis or hydrea are allowed;
5. In those patients that have received prior therapy, at least 2 weeks need to have elapsed before participating in this study. Treatment may start earlier if deemed in the best interest of the patient after discussion with the PI of the study ;
6. Eastern Cooperative Oncology Group (ECOG) performance status </= 2
7. Serum biochemical values with the following limits unless considered due to leukemia: creatinine </=2 mg/dl; total bilirubin </=2 mg/dL, unless increase is due to hemolysis or congenital disorder; transaminases (SGPT or SGOT) </=2.5* upper limit of normal (ULN);
8. Ability to swallow oral medication;
9. Ability to understand and provide signed informed consent;
10. Cardiac ejection fraction must be >/=50% (by either multiple gated acquisition scan (MUGA) scan or echocardiography).
11. Diagnosis of 1) AML (WHO classification definition of > 20% blasts), or 2) intermediate-2 or high-risk MDS (defined by the International Prognostic Scoring System (IPSS) classification) with Flt-3 mutation. Flt-3 extension phase.
12. Patients aged 15 to 65 years are eligible. Flt-3 extension phase.
13. Patients with relapsed or refractory disease or patients with secondary untreated disease are eligible, however, these patients must not have had prior exposure to a histone deacetylase inhibitor. All patients should be Flt-3 positive. Flt-3 extension phase.
14. Patients with newly diagnosed Flt3 positive AML are allowed. Flt-3 extension phase.
15. In those patients that have received prior therapy, at least 2 weeks need to have elapsed before participating in this study. Treatment may start earlier if deemed in the best interest of the patient after discussion with the PI of the study. Flt-3 extension phase.
16. ECOG performance status </= 2. Flt-3 extension phase.
17. Serum biochemical values with the following limits unless considered due to leukemia. creatinine </=2 mg/dl; total bilirubin </=2 mg/dL, unless increase is due to hemolysis or congenital disorder - transaminases (SGPT or SGOT) </=2.5* ULN. Flt-3 extension phase.
18. Ability to swallow oral medication. Flt-3 extension phase.
19. Ability to understand and provide signed informed consent. Flt-3 extension phase.
20. Cardiac ejection fraction must be >/=50% (by either MUGA scan or echocardiography). Flt-3 extension phase.

Exclusion Criteria:

1. Diagnosis of acute promyelocytic leukemia;
2. Active, uncontrolled, systemic infection considered opportunistic, life threatening or clinical significant at the time of treatment, or any severe concurrent disease, which in the opinion of the investigator and after discussion with the principal investigator, would make the patient inappropriate for study entry;
3. Male and female patients who are fertile agree to use an effective barrier method of birth control (i.e., latex condom, diaphragm, cervical cap, etc.) to avoid pregnancy. Female patients need a negative serum or urine pregnancy test within 7 days of study enrollment (applies only if patient of childbearing potential. Non childbearing is defined as 1 year or more postmenopausal or surgically sterilized);
4. Symptomatic central nervous system (CNS) involvement;
5. Patient is unable to take and/or tolerate oral medications on a continuous basis;
6. Patient has known human immunodeficiency virus (HIV) infection or known HIV-related malignancy;
7. Patient has active hepatitis B or C infection. Active disease is defined as elevated liver enzymes and/or clinical symptoms of hepatitis in addition to positive blood test for hepatitis surface antigen. In the absence of elevated liver enzymes and/or clinical symptoms, the blood test for hepatitis core antigens is not required.
8. Patient is pregnant or breast-feeding;
9. Patient has a known allergy or hypersensitivity to any component of vorinostat;
10. Patient has a history of thrombotic disorders;
11. History of any psychiatric condition that might impair the patient's ability to understand or to comply with the requirements of the study or to provide informed consent.
12. Diagnosis of acute promyelocytic leukemia. Flt-3 extension phase.
13. Active, uncontrolled, systemic infection considered opportunistic, life threatening or clinical significant at the time of treatment, or any severe concurrent disease, which in the opinion of the investigator and after discussion with the principal investigator, would make the patient inappropriate for study entry. Flt-3 extension phase.
14. Male and female patients who are fertile agree to use an effective barrier method of birth control (i.e., latex condom, diaphragm, cervical cap, etc.) to avoid pregnancy. Female patients need a negative serum or urine pregnancy test within 7 days of study enrollment (applies only if patient of childbearing potential. Non childbearing is defined as 1 year or more postmenopausal or surgically sterilized). Flt-3 extension phase.
15. Symptomatic CNS involvement. Flt-3 extension phase.
16. Patient is unable to take and/or tolerate oral medications on a continuous basis. Flt-3 extension phase.
17. Patient has known human immunodeficiency virus (HIV) infection or known HIV-related malignancy. Flt-3 extension phase.
18. Patient has active hepatitis B or C infection. Active disease is defined as elevated liver enzymes and/or clinical symptoms of hepatitis in addition to positive blood test for hepatitis surface antigen. In the absence of elevated liver enzymes and/or clinical symptoms, the blood test for hepatitis core antigens is not required. Flt-3 extension phase.
19. Patient is pregnant or breast-feeding. Flt-3 extension phase.
20. Patient has a known allergy or hypersensitivity to any component of vorinostat. Flt-3 extension phase.
21. Patient has a history of thrombotic disorders. Flt-3 extension phase.
22. History of any psychiatric condition that might impair the patient's ability to understand or to comply with the requirements of the study or to provide informed consent. Flt-3 extension phase.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2008-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, M.D., Study Chair — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center's Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Of the 106 participants enrolled, three participants completed the study's first run-in induction portion then another 103 participants were enrolled for the second portion of combined drug induction and maintenance. Four of those 103 enrolled participants were not treated.
Period: Overall Study
Arm/Group | Idarubicin + Ara-C + Vorinostat
Started | 106
Run-in Induction Phase | 3 (Initial run-in: Vorinostat induction dose 500 mg orally three times daily for 3 days.)
Induction Phase | 103 (Induction phase following determination of safe combination Vorinostat with Idarubicin.)
Completed | 99
Not Completed | 7
Not completed — Adverse Event | 1
Not completed — Death | 2
Not completed — Insurance Issues | 2
Not completed — Move to different clinical trial | 2

BASELINE CHARACTERISTICS:
Population: Three participants completed the first run-in portion of the study while 99 of remaining 103 additional participants were evaluable for the second phase of the study.
Arm/Group | Idarubicin + Ara-C + Vorinostat
Number analyzed (Participants) | 106
Age, Continuous [Median (Full Range); unit: years] | 52 [19 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 53
Region of Enrollment [Number; unit: participants]
  United States | 106

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) at 7 Months
Description: Progression-free survival defined as time from date of randomization to first occurrence of having documented disease progression or death due to any cause, whichever comes first. Progression based on tumor assessments according to Response Evaluation Criteria in Solid Tumors (RECIST). Participants were followed from baseline to disease progression with PFS evaluation at 7 months.
Time Frame: PFS Evaluation at 7 months
Population: Four (4) participants did not receive treatment therefore were not evaluable for outcome assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Idarubicin + Ara-C + Vorinostat
Number analyzed (Participants) | 102
percentage of participants | 65

2. Secondary Outcome: Participant Response
Description: Number of participants with response assessed according RECIST: Complete Response (CR) defined as normalization of marrow (< 5% blasts) and of peripheral blood counts (neutrophil count > 1.109/L, platelet count > 100 x 109/L). Partial response (PR) defined as for CR in terms of peripheral counts but with reduction of marrow blasts by >50% compared to pretreatment values but above <5%. Complete Response without platelet recovery (CRp) = CR, but platelets <100 x 109/L. Progressive disease (PD) defined as increase of blasts to > 10% after an initial response.
Time Frame: Monitoring with each 4 week cycle, up to 18 cycles of treatment
Population: Four (4) participants were not treated therefore not evaluable for the outcome assessment.
Measure: Number; unit: participants
Arm/Group | Idarubicin + Ara-C + Vorinostat
Number analyzed (Participants) | 102
participants
  Complete Response (CR) | 67
  Partial Response (PR) | 0
  Complete Response without platelet recovery (CRp) | 11
  Progressive Disease (PD) | 0
  No response | 24

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data collected while participants received study drugs up to 18 cycles (4-6 week cycles). Overall study period: 4/15/08 to 4/15/13. Four of the study's second group were not treated and therefore excluded from AE reporting.
Groups:
- Idarubicin + Ara-C + Vorinostat (Phase 1); Idarubicin + Ara-C + Vorinostat (Phase 2): Idarubicin 12 mg/m^2 by vein (IV) over 1 hour daily for 3 days (days 4 to 6). Ara-C (Cytarabine) 1.5 g/m^2 IV as a continuous infusion over 24 hours daily (days 4 to 7). Vorinostat initial dose level 500 mg orally three times a day for 3 days (days 1 to 3).
Arm/Group | Idarubicin + Ara-C + Vorinostat (Phase 1) | Idarubicin + Ara-C + Vorinostat (Phase 2)
Serious Adverse Events (participants affected / at risk) | 0/3 | 3/99
Other Adverse Events (participants affected / at risk) | 3/3 | 91/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Idarubicin + Ara-C + Vorinostat (Phase 1) (N=3) | Idarubicin + Ara-C + Vorinostat (Phase 2) (N=99)
Death (General disorders) | 0 (0) | 2 (2)
Metabolic/Laboratory, Other (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Idarubicin + Ara-C + Vorinostat (Phase 1) (N=3) | Idarubicin + Ara-C + Vorinostat (Phase 2) (N=99)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cardiac Arrhythmia-Other (Specify) (Cardiac disorders) | 0 (0) | 6 (6)
Ventricular arrhythmia--Select (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac General-Other (Specify) (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac ischemia/infarction (Cardiac disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 2 (2)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 (0) | 5 (5)
Dermatology/Skin, Other disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2) | 31 (32)
Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 71 (81)
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 1 (1) | 9 (9)
Nausea (Gastrointestinal disorders) | 2 (2) | 18 (20)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hematoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemorrhage, CNS (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hemorrhage, GI--Select (Blood and lymphatic system disorders) | 0 (0) | 5 (5)
Hemorrhage, GU--Select (Blood and lymphatic system disorders) | 0 (0) | 5 (7)
Hemorrhage/Bleeding (Blood and lymphatic system disorders) | 0 (0) | 6 (7)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Febrile neutropenia (fever unknown origin without clinical/microbiological documented infection) (Infections and infestations) | 0 (0) | 67 (111)
Infection (documented clinical/microbiologically), Grade 3-4 neutrophils (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 3 (4) | 4 (4)
Opportunistic infection associated with Grade 2 or more Lymphopenia (Infections and infestations) | 0 (0) | 29 (31)
Edema: head and neck (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Edema: limb (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Edema: trunk/genital (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
ALT, SGPT (serum glutamic pyruvic transaminase) - (Metabolism and nutrition disorders) | 0 (0) | 12 (16)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 0 (0) | 12 (13)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Mental status (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 0 (0) | 3 (3)
Scleral necrosis/melt (Eye disorders) | 0 (0) | 1 (1)
Pain-Other (General disorders) | 0 (0) | 6 (9)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes